CLINICAL TRIAL: NCT04872972
Title: Scale-up and Introduction of Simulation Into Four New Health Professional Training Institutions in East and West Africa and the Factors That Influence Simulation Adoption at These Sites
Brief Title: Scale-up the Introduction of Simulation Into Four New Health Professional Training Institutions in East and West Africa
Acronym: Sim-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other); The ELMA Foundation (Other); Alberta Children's Hospital Research Institute (Other); Laerdal Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/MUST-2/SIM-II
Record Dates: First submitted 2021-04-18; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Simulation-based Learning
Keywords: Simulation based learning

STUDY DESIGN:
Intervention Model Description: Before and After approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before/After (Other): Before and after simulation; Institutional faculty and facilities
  Interventions: Other: Simulation based learning

INTERVENTIONS:
Other: Simulation based learning — Faculty development courses on simulation based learning

SUMMARY:
Simulation based learning practice is limited in Sub-Saharan Africa. Experiences gained from our prior implementation in Phase I of this program show that simulation is feasible and significantly contributes to learning. However, the growth and sustainability of simulation methodologies in health training and service delivery institutions is subject to variability and institution specific factors. These factors may include but are not limited to ease of adoption of new technologies, human resources, space and institutional culture. These factors are likely to vary widely in Sub-Saharan Africa across countries and institutions.

It's not known how institutional factors will influence the introduction, adoption and sustainability of simulation methodologies in East and West African health training and service delivery institutions. We have partnered with four institutions in East and West Africa (in Uganda, Tanzania, and Nigeria) to learn about the process of introduction and scaling of simulation based learning in new frontiers.

DETAILED DESCRIPTION:
The investigators in this proposal have partnered and propose to expand Simulation Based Learning to Lira University in northern Uganda, Busitema University in Eastern Uganda, the Catholic University of Health and Allied Sciences (CUHAS), Tanzania and University of Jos in Nigeria. All these health training and service institutions serve large rural and peri-urban populations with poor access to health care.

The investigators will engage the partners in the co-design of implementation plans to design solutions for the barriers to implementation that are anticipated, and ensure appropriate tailoring to the local context. The investigators will use a Train of trainers (ToT) Faculty development model and this will include web-based debrief mentorship using recorded debriefing sessions from real simulations at partner sites. These videos will be loaded onto a centralization server to facilitate peer-to-peer feedback using a quality of debriefing framework.

Based on the investigators' learning experience from Phase I of implementation, the team aims to develop two categories of simulation facilitators: 1) Simulation implementation faculty (SiF) and 2) Lead simulation faculty. Lead simulation faculty (LsF) will be trained at the Mbarara University of Science and Technology (MUST) simulation center of excellence and will receive support in assessing their sites' barriers and facilitators regarding the Sim intervention. The faculty trainees will undergo an intensive 1.5-day faculty development course followed by a 2-day placement at MUST sim center for mentored scenario execution practice.

ELIGIBILITY:
Inclusion Criteria:

* Health professions Institutions in East and West Africa in the Sim for life program
* Institutional commitment to adopt simulation based learning Faculty at these health professions institutions

Exclusion Criteria: Institutions outside East and West Africa Sim for life program

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Adoption of simulation based learning | Change from baseline to 12 months after introduction of simulation based techniques
  Adoption of simulation based learning
Barriers to simulation | Change from baseline to 12 months after introduction of simulation based techniques
  Barriers to simulation based learning

SECONDARY OUTCOMES:
Facilitators | Change from baseline to 12 months after introduction of simulation based techniques
  Facilitators of simulation based learning
Institutional readiness | Change from baseline to 12 months after introduction of simulation based learning
  Institutional readiness to adopt simulation based learning

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
Ethics approval is required